CLINICAL TRIAL: NCT01441921
Title: Effect of Pistachio Intake on Insulin Resistance and Type 2 Diabetes Mellitus
Acronym: EPIRDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Western Pistachio Association (Other)
Responsible Party: Principal Investigator, Dra Monica Bullo, Principal Investigators, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PV11059S
Record Dates: First submitted 2011-09-20; First posted 2011-09-28 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: pistachio intake; insulin resistance; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control diet (Active Comparator): Low-fat normocaloric diet (30% fat, 55% carbohydrates, 15% proteins)
  Interventions: Other: control diet
- Pistachio diet (Experimental): Diet supplemented with 2 ounces of pistachio (35% fat, 50% carbohydrates adn 15% protein)
  Interventions: Dietary Supplement: Pistachios

INTERVENTIONS:
Dietary Supplement: Pistachios — Participants are randomised crossover clinical trial of 4-months trials separated by a 2-week washout period.
  Total duration of intervention and follow-up is nine months.
  Arms: Pistachio diet
Other: control diet — Participants are randomised crossover clinical trial of 4-months trials separated by a 2-week washout period.
  Total duration of intervention and follow-up is nine months.
  Arms: Control diet

SUMMARY:
Hypothesis: Chronic intake of pistachios improves glucose metabolism and insulin resistance status thus contributing to decrease the risk of type 2 diabetes mellitus and its associated abnormalities.

DETAILED DESCRIPTION:
In free-living overweight or obese adult with impaired fasting glucose or impaired glucose tolerance we will compare the effects of a pistachio-rich diet or a Mediterranean Diet on:

* Fasting glucose levels, hemoglobin A1c, insulin, C peptide, HOMA IR, advanced glycation end products and soluble receptor of advanced glycation-end products.
* Peripheral haemostatic parameters.
* Plasma inflammatory markers.
* Lymphocyte expression of toll-like receptors, C peptide, resistin and interleukin-6 in peripheral leukocytes.
* Lymphocyte glucose transport and expression of glucose transporter 4 in peripheral blood leukocytes.
* Platelet function including platelet number, mean platelet volume, platelet factor 4 levels and urinary 11-dehydro-thromboxane B2.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 35 kg/m2.
* Fasting plasma glucose levels between 100 and 125 mg/dl or
* Oral glucose tolerance test of 140 to 199 mg/dl.

Exclusion Criteria:

* Diabetes mellitus.
* Alcohol, tobacco, or drug abuse.
* Significant liver, kidney, thyroid, or other endocrine diseases.
* Frequent consumption of nuts or known history of allergy to them.
* Use of plant sterol, oral antidiabetic drugs, supplemental use of phyllium, fish oil supplements and multivitamins, vitamin E or other antioxidant supplements.
* Bad dentures, implying difficulty to chew pistachios.
* Being pregnant or wishing to become a pregnant 6 months before or during the study, lactating 6wk before or during the study.
* Following vegetarian or weight loss diets.
* Other medical or social conditions that difficult the compliance to the intervention.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in circulating levels of glucose and insulin according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  Measurement of circulating glucose and insulin levels and cellular glucose uptake

SECONDARY OUTCOMES:
Changes from baseline in inflammatory, oxidative and metabolic risk markers related to glucose/insulin metabolism according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  Cpeptide, resistin, IL-6, IL-18, Ghrelin, leptin, adiponectin, GLP-1 and oxidized LDL will be measured.
Changes from baseline in haemostatic parameters according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  Tissue factor, fibrinogen, PAI-1, vWF will be measured.
Changes from baseline in HL and LDL size according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  Plasmi lipoprotein size will be measured by polycacrylamide gradient gel electrophoresis
Changes in advanced glycation end products according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  Advanced glycation end products and soluble receptor of advanced glycation-end produtcs will be measured
Changes from baseline in gene expression in the peripheral cells according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  RNA from peripheral leukocytes will be isolated for the subsequent measurements of changes in gene expression of toll-like receptors, GLUT-4, C-peptide, resistin adn IL-6, and genes involved in telomere maintenance and oxidation
Changes from baseline in cellular glucose uptake according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  Glucose uptake and GLUT4 protein levels will be assessed in peripheral leukocytes
Changes from baseline in platelet function according to the intervention arm | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first and second intervention arm
  Platelet number, mean platelet volume and platelet factor 4 in blood, and urinary levels of 11-dehydro-thromboxane B2 will be assessed.
Changes from baseline in telomeric length of leukocytes (LTL) | Participants will be followed for 9 months. Measurements will be done before and after 4 months of the first intervention arm. Measurements will be not analysed after the second period due to expected carry-over effect.
  Telomere lenght will be evaluated as a biomarker of biological age and general health status. Telomere attrition may play an important role in the pathogenesis and severity of type 2 diabetes (T2D) increasing the probability of beta-cell senescence, leading to reduced cell mass and decreased insulin secretion.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bullo, Dra., Principal Investigator — Institut Investigacio Sanitaria Pere Virgili
Locations (1):
- Human Nutrition Unit, Faculty of Medicine, Rovira i Virgili University, Reus, Tarragona, Spain

REFERENCES:
- [Background] Hernandez-Alonso P, Salas-Salvado J, Baldrich-Mora M, Mallol R, Correig X, Bullo M. Effect of pistachio consumption on plasma lipoprotein subclasses in pre-diabetic subjects. Nutr Metab Cardiovasc Dis. 2015 Apr;25(4):396-402. doi: 10.1016/j.numecd.2015.01.013. Epub 2015 Feb 7. PMID 25791863
- [Result] Hernandez-Alonso P, Salas-Salvado J, Baldrich-Mora M, Juanola-Falgarona M, Bullo M. Beneficial effect of pistachio consumption on glucose metabolism, insulin resistance, inflammation, and related metabolic risk markers: a randomized clinical trial. Diabetes Care. 2014 Nov;37(11):3098-105. doi: 10.2337/dc14-1431. Epub 2014 Aug 14. PMID 25125505
- [Result] Hernandez-Alonso P, Canueto D, Giardina S, Salas-Salvado J, Canellas N, Correig X, Bullo M. Effect of pistachio consumption on the modulation of urinary gut microbiota-related metabolites in prediabetic subjects. J Nutr Biochem. 2017 Jul;45:48-53. doi: 10.1016/j.jnutbio.2017.04.002. Epub 2017 Apr 12. PMID 28432876
- [Result] Hernandez-Alonso P, Giardina S, Salas-Salvado J, Arcelin P, Bullo M. Chronic pistachio intake modulates circulating microRNAs related to glucose metabolism and insulin resistance in prediabetic subjects. Eur J Nutr. 2017 Sep;56(6):2181-2191. doi: 10.1007/s00394-016-1262-5. Epub 2016 Jul 6. PMID 27383196
- [Derived] Canudas S, Hernandez-Alonso P, Galie S, Muralidharan J, Morell-Azanza L, Zalba G, Garcia-Gavilan J, Marti A, Salas-Salvado J, Bullo M. Pistachio consumption modulates DNA oxidation and genes related to telomere maintenance: a crossover randomized clinical trial. Am J Clin Nutr. 2019 Jun 1;109(6):1738-1745. doi: 10.1093/ajcn/nqz048. PMID 31051499
- See also: Related Info — http://www.iispv.cat/